CLINICAL TRIAL: NCT06710119
Title: Effect of Custom Dynamic Orthoses on Forefoot Loading
Acronym: LoadsolCP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iowa (Other)
Collaborators: Cornerstone Clinics, Everett, WA (Unknown)
Responsible Party: Principal Investigator, Jason Wilken, Associate Professor, University of Iowa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 202207100
Record Dates: First submitted 2024-11-25; First posted 2024-11-29 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Lower Extremity Injuries
Keywords: Gait Analysis; Ankle Foot Orthosis; Carbon Fiber; Biomechanics; Visual Feedback; Foot Loading
MeSH Terms: interventions — Feedback, Sensory

STUDY DESIGN:
Intervention Model Description: Participants will either receive training with or without visual feedback of foot loading during gait.
Masking Description: Participants will not be blinded to which study arm they are assigned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- No Visual Feedback (No Intervention): Participants will receive typical accommodation training after being prescribed the CDO.
- Provided Visual Feedback (Active Comparator): Participants will receive typical accommodation training with additional visual feedback after being prescribed the CDO.
  Interventions: Other: Visual Feedback

INTERVENTIONS:
Other: Visual Feedback — Visual feedback of foot loading during gait.
  Arms: Provided Visual Feedback

SUMMARY:
The proposed study is designed to evaluate how foot loading changes during initial accommodation to a carbon fiber custom dynamic orthosis (CDO), after targeted training with or without visual feedback of foot loading, and after take-home use of the CDO. This study will quantify initial offloading associated with CDO use and determine if visual feedback of foot loading and additional take-home use of the CDO can further reduce forces, as orthotists work to provide CDOs to patients.

DETAILED DESCRIPTION:
This study is designed to evaluate the effects of initial accommodation, CDO related training, and take-home use on foot loading during gait. In this study, adult participants who experienced an injury below the knee and require a CDO will walk without the CDO, then with the CDO following initial prescription, after training with or without visual force feedback, and after additional take-home use of the CDO. Participants will be randomized to to training with or without visual feedback of foot loading forces.

Wireless force measuring sensors will be used to measure forces under the foot with and without the CDO at each time point. Participants will complete questionnaires to assess and compare various patient outcomes (e.g. pain, quality of life, comfort, satisfaction, and preference).

ELIGIBILITY:
Patient Inclusion criteria

* Ages: 18-65
* Sustained a function limiting injury below the knee, requiring a carbon fiber custom dynamic orthosis
* Shoe size between women's 8 and 13.5 or men's 6.5 and 13
* Any of the following: weakness of ankle plantarflexors (<4/5 on MMT), limited pain free ankle motion (DF<10deg or PF<20deg), mechanical pain with loading onto hindfoot/midfoot/forefoot (>4/10 on verbal numeric pain rating scale), ankle or hindfoot fusion, candidate for ankle or hindfoot fusion, candidate for amputation secondary to ankle/foot impairment
* Ability to walk 25 feet without using a cane or crutch
* Ability to walk at a slow to moderate pace
* Able to read and write in English and provide written informed consent

Patient Exclusion criteria

* Pain > 9/10 while walking
* Ankle weakness as a result of spinal cord injury or central nervous system pathology
* AFO or CDO prescription that includes a knee brace or goes up to thigh
* Medical or psychological conditions that would preclude functional testing (ex. severe traumatic brain injury, heart condition, clotting disorder, lung condition, stroke, vestibular disorder)
* Nerve, muscle, bone, or other condition limiting function of the contralateral extremity
* BMI greater than 40
* Visual or hearing impairment that limit walking ability or limit the ability to comply with instructions given during testing
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06-18 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Peak Plantar Force (Forefoot) | Baseline
  Maximum force (N) collected from the forefoot (distal 40% of sensor) during gait.
Plantar Force Impulse (Forefoot) | Baseline
  Plantar force impulse (Ns) across the forefoot (distal 40% of sensor) will be calculated using the integral of the force over the stance phase as participants walk.

SECONDARY OUTCOMES:
Peak Plantar Force (Midfoot) | Baseline
  Maximum force (N) collected from the midfoot (middle 30% of sensor) during gait.
Plantar Force Impulse (Midfoot) | Baseline
  Plantar force impulse (Ns) across the midfoot (middle 30% of sensor) will be calculated using the integral of the force over the stance phase as participants walk.
Peak Plantar Force (Hindfoot) | Baseline
  Maximum force (N) collected from the hindfoot (proximal 30% of sensor) during gait.
Plantar Force Impulse (Hindfoot) | Baseline
  Plantar force impulse (Ns) across the hindfoot (proximal 30% of sensor) will be calculated using the integral of the force over the stance phase as participants walk.
Peak Plantar Force (Total Foot) | Baseline
  Maximum force (N) collected from the total foot (100% of sensor) during gait.
Plantar Force Impulse (Total Foot) | Baseline
  Plantar force impulse (Ns) across the total foot (100% of sensor) will be calculated using the integral of the force over the stance phase as participants walk.

OTHER OUTCOMES:
Modified Socket Comfort Score (Comfort) | Baseline
  Comfort scores range from 0 = most uncomfortable to 10 = most comfortable.
Modified Socket Comfort Score (Smoothness) | Baseline
  Smoothness scores range from 0 = least smooth to 10 = most smooth.
Numerical Pain Rating Scale | Baseline
  Pain will be assessed using a standard 11-point numerical pain rating scale, in which 0 = no pain and 10 = worst pain imaginable.
Patient Reported Outcome Measurement Information System (Physical Function) | Baseline
  The Patient Reported Outcome Information System (PROMIS) physical function Computer Adaptive Test (CAT) is a computerized assessment measuring physical function. It is scored using a T-score in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population. In a given PROMIS domain, a T-score above 50 represents more of the measured variable than the population average.
Patient Reported Outcome Measurement Information System (Pain Interference) | Baseline
  The Patient Reported Outcome Information System (PROMIS) pain interference Computer Adaptive Test (CAT) is a computerized assessment measuring pain interference. It is scored using a T-score in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population. In a given PROMIS domain, a T-score above 50 represents more of the measured variable than the population average.
Orthotics and Prosthetics User Survey - Satisfaction with Service | Baseline
  Satisfaction with services will be assessed using the Orthotics Prosthetics Users' Survey Satisfaction With Services Score (10-50). Lower scores indicate a better outcome.
Orthotics and Prosthetics User Survey - Satisfaction with Device | Baseline
  Satisfaction with device will be assessed using the Orthotics Prosthetics Users' Survey Satisfaction With Device Score (11-55). Lower scores indicate a better outcome.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Iowa, Iowa City, Iowa
  - Cornerstone Prosthetics and Orthotics, Everett, Washington

IPD SHARING:
Plan to Share IPD: No